CLINICAL TRIAL: NCT00397137
Title: Prospective Randomized Multi-centre Trial Comparing the Clinical Efficacy, Safety and Patient Acceptability of Circular Stapled Anopexy With Closed Diathermy Haemorrhoidectomy for Haemorrhoids
Brief Title: Stapled Anopexy Versus Closed Haemorrhoidectomy for Haemorrhoids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Ethicon Endo-Surgery (Industry); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202/99
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Hemorrhoids
Keywords: Symptomatic haemorrhoids; haemorrhoidectomy; stapled anopexy
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stapled Anopexy (Experimental): Circular stapled anopexy
  Interventions: Procedure: Circular stapled anopexy
- Conventional Haemorrhoidectomy (Active Comparator): Closed diathermy haemorrhoidectomy
  Interventions: Procedure: Closed diathermy haemorrhoidectomy

INTERVENTIONS:
Procedure: Circular stapled anopexy — Patients receiving stapled anopexy to treat haemorrhoids
  Arms: Stapled Anopexy
Procedure: Closed diathermy haemorrhoidectomy — Conventional haemorrhoidectomy as described by Ferguson method
  Arms: Conventional Haemorrhoidectomy

SUMMARY:
The aim of this study is to determine the role of stapled anopexy in the treatment of haemorrhoids by comparing it to the current gold standard treatment, which is excisional haemorrhoidectomy.

DETAILED DESCRIPTION:
The current gold standard treatment of haemorrhoids namely, excisional haemorrhoidectomy is associated with severe postoperative pain and prolonged recovery period. Methods aiming at improving the outcome of excisional surgery included mainly modifications of the existing technique. Alternative instruments other than scissors have been used for the actual excision of haemorrhoids with a view to reducing the postoperative pain. However, with the wound in the sensitive anoderm following excisional haemorrhoidectomy, pain continues to be a major problem irrespective of the method of excision or of the instrument employed.

The new technique of stapled anopexy introduced in 1998 uses a radically different approach to treat haemorrhoids. The prolapsed anal cushion is repositioned and fixed without actually excising the haemorrhoidal pedicle thereby avoiding an external wound. This should result in reduction of the postoperative pain and subsequently should improve the recovery time. Further potential advantages of the technique should include a more physiological approach to the treatment of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult human subjects (age >=16 years) with symptomatic haemorrhoids (Primary or recurrent)
* symptomatic haemorrhoids (grades 2, 3, 4) needing surgical treatment

Exclusion Criteria:

* concurrent untreated or recurrent colorectal cancer
* Active inflammatory bowel disease
* Previous major anorectal surgery
* On anticoagulant medications
* Non-consenting patients
* Unwilling for randomisation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2000-09; Primary Completion 2003-10 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain
global haemorrhoidal symptom control
complication rates

SECONDARY OUTCOMES:
Time to recovery
Time to return to work
Re-treatment rates
Day case surgeries
Quality of life changes
Patient satisfaction
Cost effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Robert JC Steele, MD, Principal Investigator — University of Dundee; Mohamed A Thaha, MRCS, Principal Investigator — University of Dundee
Locations (1):
- Ninewells Hospital & Medical School, Dundee, Scotland, United Kingdom

REFERENCES:
- [Result] Thaha MA, Irvine LA, Steele RJ, Campbell KL. Postdefaecation pain syndrome after circular stapled anopexy is abolished by oral nifedipine. Br J Surg. 2005 Feb;92(2):208-10. doi: 10.1002/bjs.4773. PMID 15584064
- [Result] Thaha MA, Campbell KL, Kazmi SA, Irvine LA, Khalil A, Binnie NR, Hendry WS, Walker A, Staines HJ, Steele RJ. Prospective randomised multi-centre trial comparing the clinical efficacy, safety and patient acceptability of circular stapled anopexy with closed diathermy haemorrhoidectomy. Gut. 2009 May;58(5):668-78. doi: 10.1136/gut.2008.151266. Epub 2008 Dec 17. PMID 19091821